CLINICAL TRIAL: NCT02184767
Title: A Nonrandomized, Open-Label, Multicenter, Phase 1 Study to Assess the Safety and Pharmacokinetics of ADASUVE® (STACCATO® Loxapine for Inhalation) at Doses of 2.5, 5, or 10 mg in Children and Adolescents (10 Through 17 Years of Age) With Any Condition Warranting Chronic Use of an Antipsychotic Medication
Brief Title: Study to Assess the Safety and Pharmacokinetics of ADASUVE® at Doses of 2.5, 5, or 10 mg in Children and Adolescents (10 Through 17 Years of Age) With Any Condition Warranting Chronic Use of an Antipsychotic Medication
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TV571-CNS-10018
Record Dates: First submitted 2014-07-03; First posted 2014-07-09 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: BiPolar
MeSH Terms: interventions — Loxapine; Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADASUVE® (Experimental): oral inhalation using a single-use, hand-held, inhaler; dosage determined by the investigator according the participants weight
  Interventions: Drug: ADASUVE®

INTERVENTIONS:
Drug: ADASUVE® — ADASUVE® 2.5, 5, or 10 mg
  Other Names: STACCATO® Loxapine for Inhalation

SUMMARY:
This study is to assess the pharmacokinetics of loxapine and will be using plasma concentration data obtained over 48 hours after administration of the study drug

ELIGIBILITY:
Inclusion

1. Written informed consent is obtained from each patient's parent or legal guardian and written assent is obtained from each patient.
2. The patient is a boy or girl 10 through 17 years of age.
3. The patient is within the 2.5 to 97.5 percentile for body mass index (BMI) on the basis of age and sex and is within the following weight range, as appropriate:

   * boys: more than 27 kg and 127 kg or less
   * girls: more than 27 kg and 111 kg or less
4. The patient has a documented history of schizophrenia, bipolar disorder, autism, or any condition for which the use of antipsychotic medication (eg, risperidone, olanzapine, aripirazole, haloperidol, etc.) is warranted and/or administered. Note: Patients currently receiving treatment for any condition must be on a stable regimen (dose and frequency) for a minimum of 28 days before administration of ADASUVE.
5. The patient is in good general health as determined by a complete medical history (including psychiatric and respiratory), clinical laboratory tests (include hematology, serum chemistry, and urinalysis), physical examination, body weight, 12-lead ECG, spirometry, vital signs measurements (blood pressure [systolic and diastolic], heart rate, body temperature, and respiratory rate), pulse oximetry, chest auscultation, neurologic examination, suicidality assessment, and concomitant medication usage inquiry.
6. Female patients who are postmenarche or sexually active must have a negative pregnancy test result, must have exclusively same sex partners or be using an acceptable method of contraception, and must agree to continued use of this method for the duration of the study and for 30 days after discontinuation of ADASUVE. Acceptable methods of contraception include abstinence or an intrauterine device (known to have a failure rate of less than 1% per year).
7. The patient has negative alcohol test and urine drug screen (UDS) results. A positive UDS result with appropriate medical explanation (eg, prescribed amphetamines) may be permitted after consultation with the medical monitor. Note: The UDS will also detect the presence of tetrahydrocannabinol (THC). A positive result for THC may be permitted after discussion with the sponsor if the result is low and is consistent (eg, positive at all predose assessments). If a patient tests negative for THC at screening, the result must remain negative at check-in for the patient to be eligible for study participation.
8. The patient and parent/legal guardian must be willing and able to comply with study restrictions and to remain at the investigational center for the required duration at each visit.

Exclusion

1. The patient has any clinically significant uncontrolled medical condition (treated or untreated) other than the conditions specified in inclusion criterion d.
2. The patient has a current diagnosis or history of asthma, chronic obstructive pulmonary disease (COPD), bronchiolitis, chronic bronchitis, emphysema, or other lung disease associated with bronchospasm.
3. The patient has acute respiratory signs or symptoms (eg, wheezing)
4. The patient currently has or has a known history of the following:

   * cardiovascular disease (including, but not limited to, myocardial infarction or ischemic heart disease, heart failure, or conduction abnormalities)
   * cerebrovascular disease
   * conditions that predispose him or her to hypotension (including, but not limited to, dehydration, hypovolemia, or treatment with antihypertensive medications or other drugs that affect blood pressure or reduce heart rate)
   * seizure disorder except a history of infantile febrile seizures
5. The patient is pregnant or lactating.
6. The patient is febrile.
7. The patient has any other disease or condition that, in the investigator's or medical monitor's opinion, would present undue risk to the patient, or may confound the interpretation of study results.
8. The patient has taken any of the following drugs, substances, or foods:

   * any investigational drug within 30 days or 5 half-lives (whichever is longer) before administration of ADASUVE or, in the case of a new chemical entity, 3 months or 5 half-lives (whichever is longer) before administration of ADASUVE
   * current use of medications to treat airway disease such as asthma or COPD
   * loxapine or amoxapine within the last 30 days
   * more than 21 units of alcohol per week within the past 2 years or a history of alcohol, narcotic, or any other substance abuse or dependence as defined by the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR, American Psychiatric Association 2000). Note: A unit of alcohol is equal to 1 ounce of hard liquor, 5 ounces of wine, or 8 ounces of beer.
   * clinically significant excessive consumption of coffee, tea, and/or other caffeine-containing beverage or food (ie, 600 mg of caffeine or more per day, or 12-ounce caffeine-containing sodas, 30 ounces of chocolate, or 5 or more cups of coffee per day), or a combination of any of these beverages or foods within 2 weeks before the dose of ADASUVE
   * nicotine-containing products (including but not limited to cigarettes, cigars, and chewing or dipping tobacco) within 12 months before administration of ADASUVE or use of topical or oral nicotine preparations for smoking cessation within the past 3 months before administration of ADASUVE
9. The patient has a known sensitivity or idiosyncratic reaction to loxapine or amoxapine, any compound present in the study formulation, any metabolites, or any other related compounds.
10. The patient has a history of any clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, including multiple allergies or drug reactions.
11. The patient has a known history of contraindications to anticholinergics (eg, bowel obstructions, urinary retention, or acute glaucoma).
12. The patient has any procedure or disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery; a history of appendectomy is allowed).
13. The patient has received or donated blood or blood products (eg, plasma or platelets) in the 3 months before administration of ADASUVE or has made more than 2 blood (≥ 450 mL) or blood product donations within the 12 months before administration of ADASUVE, or has plans to donate during the study or within 3 months after completion of the study.
14. The patient has 1 or more clinical laboratory test values outside the range specified below, or any other clinically significant laboratory abnormality, as determined by the investigator or medical monitor:

    * hemoglobin value of less than 11.0 g/dL
    * more than twice the upper limit of the normal range (ULN)
    * total bilirubin value of more than the ULN
15. With the exception of the conditions specified in inclusion criterion d, the patient has had, within 4 weeks before administration of ADASUVE, a clinically significant illness or, within 1 week before administration of ADASUVE, has had any acute illness, or at screening or on the day before administration of ADASUVE, has symptoms of any clinically significant or acute illness.
16. The patient has a positive test result for hepatitis B surface antigen (HBsAg) or antibodies to hepatitis C virus, or has a known positive human immunodeficiency virus (HIV) history.
17. The patient is unable to tolerate direct venipuncture.
18. The patient has blood pressure outside the range of 90 to 140 mm Hg (systolic) or 50 to 90 mm Hg (diastolic). Note: Only 2 rechecks are permissible for study eligibility purposes.
19. The patient has, after resting for 5 minutes, an oxygen saturation at less than 95%. Note: Only 2 rechecks are permissible for study eligibility purposes.
20. The patient has evidence of a clinically significant ECG abnormality.
21. The patient has a forced expiratory volume in 1 second (FEV1) of less than 80% of predicted value on spirometry.
22. The patient is unlikely to comply with the study protocol, or is unsuitable for any other reasons, as judged by the investigator.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUC0-t) | 48 hours

SECONDARY OUTCOMES:
area under the plasma concentration-time curve from time 0 to infinity (AUC0-inf) | 48 hours
ratio of AUC0-t to AUC0-inf (AUC0-t/AUC0-inf) | 48 hours
maximum observed plasma drug concentration (Cmax) | 48 hours
time to maximum observed concentration (tmax) | 48 hours
apparent terminal elimination rate constant (Kel) | 48 hours
elimination half-life (t½) | 48 hours
apparent clearance (CL/F) | 48 hours
volume of distribution (V/F) | 48 hours
The palatability of ADASUVE will be performed using a visual analog scale (VAS) | 2 1/2 weeks
Summary of participants with adverse events | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (2):
- United States (2):
  - Teva Investigational Site 12468, Atlanta, Georgia
  - Teva Investigational Site 12469, Cincinnati, Ohio

REFERENCES:
- [Derived] Dong M, Fukuda T, Selim S, Smith MA, Rabinovich-Guilatt L, Cassella JV, Vinks AA. Clinical Trial Simulations and Pharmacometric Analysis in Pediatrics: Application to Inhaled Loxapine in Children and Adolescents. Clin Pharmacokinet. 2017 Oct;56(10):1207-1217. doi: 10.1007/s40262-017-0512-x. PMID 28205038